CLINICAL TRIAL: NCT02973542
Title: Evaluation of the Efficacy and Tolerance of Ethosuximide in the Treatment of Abdominal Pain Associated With Irritable Bowel Syndrome
Brief Title: Ethosuximide to Treat IBS
Acronym: IBSET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: SFETD (Socièté Française d'Etude et de Traitement de la Douleur) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-289; 2016-002110-42 (Other: 2016-002110-42)
Record Dates: First submitted 2016-11-18; First posted 2016-11-25 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2022-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Ethosuximide; Pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Pain | interventions — Ethosuximide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ethosuximide (Experimental): A responder will correspond to a decrease in abdominal pain score (11-points NRS pain) of at least 30% compared to the score before treatment and a score of 6 or 7 on the SGA scale. At endpoint (12-weeks treatment period), it will be compared the responder rate between the 2 treatment arms (ethosuximide vs placebo).
  Interventions: Drug: Ethosuximide
- placebo (Placebo Comparator): A responder will correspond to a decrease in abdominal pain score (11-points NRS pain) of at least 30% compared to the score before treatment and a score of 6 or 7 on the SGA scale. At endpoint (12-weeks treatment period), it will be compared the responder rate between the 2 treatment arms (ethosuximide vs placebo).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ethosuximide — The study will aim to evaluate the effectiveness of ethosuximide on abdominal pain in patients with IBS, its tolerance and its impact on patient quality of life, severity of symptoms related to IBS and the use of analgesics / antispasmodic / regulators transit.
  Arms: ethosuximide
Other: Placebo — The study will aim to evaluate the effectiveness of ethosuximide on abdominal pain in patients with IBS, its tolerance and its impact on patient quality of life, severity of symptoms related to IBS and the use of analgesics / antispasmodic / regulators transit.
  Arms: placebo

SUMMARY:
Abdominal pain remains the most deleterious symptom for patients with irritable bowel syndrome (IBS) and is causing a significant alteration of their quality of life. The visceral hypersensitivity seems to be one of the key mechanisms that could explain the abdominal pain in these patients. Current treatments, mainly symptomatic, are of limited effectiveness, especially in terms of relief of abdominal pain. The study will aim to evaluate the effectiveness of ethosuximide on abdominal pain in patients with IBS, its tolerance and its impact on patient quality of life, severity of symptoms related to IBS and the use of analgesics / antispasmodic / regulators transit.

DETAILED DESCRIPTION:
The irritable bowel syndrome (IBS) is characterized by a combination of discomfort and / or abdominal pain and bowel habits in the absence of identifiable organic pathology. This condition is extremely common because it is the first cause of consultation in gastroenterology and would cover 10-15% of the French. This chronic condition, although functional, impact significantly on the quality of life of patients and causes considerable health spending, making it a major public health problem. Especially as the currently used treatments are of limited effectiveness.

Among the pathophysiological mechanisms involved in IBS, visceral hypersensitivity (VHS) seems to be a major factor causing pain in patients. VHS involves sensitization of colonic nerve fibers, resulting in an increase of neuronal excitability. In several animal models of chronic pain, this hyperexcitability was related to a change in the expression or activity of ion channels, including calcium channel Cav3.2.

Investigators especially shown the involvement of Cav3.2 channels in visceral pain in an animal model of VHS. Furthermore, overexpression of these channels at the peripheral level (dorsal root ganglion innervating the colon) has been demonstrated in this animal model and pharmacological blockade, including ethosuximide, prevented the development of the VHS. Note that Cav3.2 channels have been widely demonstrated as involved in nociceptive phenomena in various animal models of chronic pain and that by blocking their ethosuximide induce an analgesic effect in these models.

Finally, we have recently demonstrated the involvement of Cav3.2 channel in patients with IBS, in a clinical case-control study. The Cav3.2 channels were overexpressed in the colonic mucosa of patients with IBS compared to asymptomatic controls.

The Cav3.2 channels are therefore a potential pharmacological target and ethosuximide a promising therapy to effectively treat the abdominal pain associated with IBS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,

  * Man,
  * Women, Negative pregnancy test and effective contraception,
  * IBS defined by the Rome criteria IV
  * During the previous seven days the inclusion visit, average NRS pain ≥ 4,
  * IBS Treatment stable for 1 month
  * Patients affiliated to the French Social Security,
  * Patients with the informed consent were obtained.

Exclusion Criteria:

* Breastfeeding
* Diabetic patients
* Known renal or hepatic impairment,
* Significant liver function abnormalities (transaminases> 3N, cholestasis) and renal (MDRD <60 ml / min)
* Addiction to alcohol and / or drugs,
* AEDs taken (epilepsy or chronic pain)
* chronic pain of greater intensity than that related to IBS,
* Allergy succinimides (ethosuximide, methsuximide, phensuximide)
* History or current severe depression (hospitalization, long-term antidepressant treatment)
* Psychotic disorders,
* Patients exclusion period, or total exceeded authorized allowances
* Patients undergoing a measure of legal protection (trusteeship, guardianship ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
30% reduction in abdominal pain | through study completion, an average of 12 weeks.
Score of 4 or 5 on the SGA scale | through study completion, an average of 12 weeks.

SECONDARY OUTCOMES:
Monthly assessment of abdominal pain | at 1 month
Monthly assessment of score of Bristol scale | at 1 month
Monthly evaluation of GIQLI questionnaire | at 1 month
Monthly evaluation of EQ-5D questionnaire | at 1 month
Monthly evaluation of IBS-SSS questionnaire | at 1 month
Monthly evaluation of SGA scale. | at 1 month
Monthly evaluation of the use of analgesics | at 1 month
Monthly evaluation of the use of antispasmodic | at 1 month
Monthly evaluation of the use of regulators transit. | at 1 month
Monthly evaluation of medical response rate | at 1 month
Monthly evaluation of stop work related to IBS. | at 1 month
Evaluation of the tolerance of ethosuximide throughout the study. | at 1 month
Evaluation of the discontinuation rate study because of adverse events throughout the study | at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Julien SCANZI, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Kerckhove N, Zerbib F, Chambaz M, Mion F, Zalar A, Goutorbe F, Coffin B, Payen L, Roman S, Guilngar A, Pereira B, Duale C, Dapoigny M, Melchior C, Scanzi J; IBSET Investigator Group (IIG). Ethosuximide and Irritable Bowel Syndrome-Related Abdominal Pain: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2551368. doi: 10.1001/jamanetworkopen.2025.51368. PMID 41505133
- [Derived] Kerckhove N, Scanzi J, Pereira B, Ardid D, Dapoigny M. Assessment of the effectiveness and safety of ethosuximide in the treatment of abdominal pain related to irritable bowel syndrome - IBSET: protocol of a randomised, parallel, controlled, double-blind and multicentre trial. BMJ Open. 2017 Jul 18;7(7):e015380. doi: 10.1136/bmjopen-2016-015380. PMID 28720615